CLINICAL TRIAL: NCT03513341
Title: Levels of Daily Physical Activity and Sedentary Behaviour in Maastricht University's Undergraduate First Year Students
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, H.Q. Chim, PhD student, Maastricht University
Other Study IDs: 808
Record Dates: First submitted 2018-03-17; First posted 2018-05-01 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Physical Activity; Sedentary Lifestyle
Keywords: Physical activity; Sedentary behaviour; Undergraduate
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maastricht University First Year Students: Maastricht University 2017-2018 undergraduate first year students are invited to participate in the study. The participants are invited to complete a demographics questionnaire, wear an ActivPAL accelerometer for 7 days, and to complete daily diaries (modified International Physical Activity Questionnaire) for 7 days.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is given to the participants. This is an observational study exploring the students' levels of physical activity and sedentary behaviour in their natural setting.

SUMMARY:
This study explores the levels of daily physical activity and sedentary behaviour in Maastricht University's undergraduate first year students. Furthermore, this study explores the correlations between the students' demographical background information with their levels of physical activity and sedentary behaviour.

DETAILED DESCRIPTION:
Participants are randomly recruited from the student population. The participants are invited to complete a demographics questionnaire, wear an ActivPAl accelerometer for 7 days, and complete daily diaries (modified International Physical Activity Questionnaire) throughout the 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Matriculated Maastricht University 2017-2018 First Year Student

Exclusion Criteria:

* Student of Maastricht University's Maastricht Science Programme (MSP) course. This is because the MSP students are undergoing another intervention (i.e., long term use of standing desks) introduced by the same team of researchers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Maastricht University 2017-2018 First Year Students
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) measured by the ActivPAL accelerometer | 7 days
  The ActivPAL accelerometer senses limb position and activity. From this information, it can reliably discriminate periods of upright activity from seated or lying activities. Furthermore, the cadence (stepping rate) of upright activities can be accurately recorded. Energy expenditure (estimated by the ActivPAL accelerometer using Metabolic Equivalent of Task (MET)) and cadence (step frequency, i.e., steps per minute) will be used to distinguish between sleeping, being sedentary, standing and stepping. The time spent sleeping, being sedentary, standing and stepping will be measured and compared against global recommendations of physical activity (e.g., WHO recommendations).

SECONDARY OUTCOMES:
Correlations (r) between age (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between age (days/months/years) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between gender (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between gender ("gender variant/non-conforming" or "male" or "female" or "transgender male" or "transgender female" or "prefer not to answer" or "not listed (please specify)") and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between height (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between height (metres) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between weight (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between weight (kilograms) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between race/ethnicity (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between race/ethnicity ("White/Caucasian" or "African" or "Middle Eastern" or "South Asian" or "Latino/Hispanic" or "East Asian" or "Caribbean" or "Prefer not to answer" or "Other (please specify)") and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between nationality (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between nationality (reported by name of nationality) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between living area (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between living area (coded as "rural" or "urban" by analysing postal code) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between education status (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between education status (years of study, years in tertiary education and hours of classes per day) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between commuting status (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between commuting status (i.e., mode of transportation, availability of transportation type, and travel duration in minutes) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between employment status (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between employment status (absence or presence of a part-time job secondary to being a student) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between living status (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between living status ("Alone", "With parent(s)/guardian(s)", "With siblings", "With friend(s)/flatmate(s)", "With partner(s)", "With child(ren)", and/or "Other (please specify)") and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between social class (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between social class (measured by the highest achieved level of education by parents(s)/guardian(s)) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between gym or sports club membership (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between gym membership (absence, presence or presence but inactive of a gym or sports club membership) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between sleep duration (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between sleep duration (hours) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between smoking status (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between smoking status ("Yes", "No, I stopped less than 6 months ago", "No, I stopped more than 6 months ago", or "No, I have never smoked") and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between smoking type (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between smoking type ("Pipe", "Cigarettes/Shag", "Cigar", "E-cigarettes/Vaporizers or any other electronic devices", "Not applicable" or "Other (please specify)") and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between smoking frequency (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between smoking frequency (counts per day) and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).
Correlations (r) between alcohol consumption (measured with a Demographics Questionnaire) and time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping; measured by the ActivPAL accelerometer) | 7 days
  The correlations between alcohol consumption ("Every day", "3-5 times a week", "Once a week", "Only on weekends", "Only on special occasions" or "Never") and the time (minutes) spent in various activities (sleeping, being sedentary, standing and stepping) will be measured to explore the determinants of the various activities (sleeping, being sedentary, standing and stepping).

CONTACTS AND LOCATIONS:
Overall Officials: Hui Qing Chim, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: A maximum of 1 year after publication of study in a journal.

REFERENCES:
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Duvivier BM, Schaper NC, Bremers MA, van Crombrugge G, Menheere PP, Kars M, Savelberg HH. Minimal intensity physical activity (standing and walking) of longer duration improves insulin action and plasma lipids more than shorter periods of moderate to vigorous exercise (cycling) in sedentary subjects when energy expenditure is comparable. PLoS One. 2013;8(2):e55542. doi: 10.1371/journal.pone.0055542. Epub 2013 Feb 13. PMID 23418444
- [Background] Penedo FJ, Dahn JR. Exercise and well-being: a review of mental and physical health benefits associated with physical activity. Curr Opin Psychiatry. 2005 Mar;18(2):189-93. doi: 10.1097/00001504-200503000-00013. PMID 16639173
- [Background] Wilmot EG, Edwardson CL, Achana FA, Davies MJ, Gorely T, Gray LJ, Khunti K, Yates T, Biddle SJ. Sedentary time in adults and the association with diabetes, cardiovascular disease and death: systematic review and meta-analysis. Diabetologia. 2012 Nov;55(11):2895-905. doi: 10.1007/s00125-012-2677-z. Epub 2012 Aug 14. PMID 22890825